CLINICAL TRIAL: NCT00241410
Title: Investigation of the Safety, Immunological Effect and Efficacy of the Combined Application of MPL and Grass Pollen Allergen
Brief Title: Safety, Immunological Effect and Efficacy of the Combined Application of MPL and Grass Pollen Allergen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Jutta Amersdorffer, Allergy Therapeutics (UK) Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OralvacB2MPL103; EudraCT No.: 2005-004095-20
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-09

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Sublingual Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4 consecutive groups, dose escalation
  Interventions: Biological: OralvacB2MPL
- 2 (Placebo Comparator): 4 consecutive groups
  Interventions: Biological: OralvacB2MPL

INTERVENTIONS:
Biological: OralvacB2MPL — Comparison of different dosages of drug
  Other Names: MPL and/or grass pollen allergen

SUMMARY:
Safety and tolerability of different dose combinations of MPL and grass pollen allergen and to identify the highest combinations of MPL and grass pollen allergen which is safe.

Pharmacodynamics and efficacy of MPL and grass pollen allergen.

DETAILED DESCRIPTION:
Objective of this trial is to demonstrate the safety and tolerability of different dose combinations of MPL and grass pollen allergen and to identify the highest combination of MPL and grass pollen allergen which is safe.

Other objectives are to investigate the pharmacodynamics and efficacy of MPL and grass pollen allergen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, between 18 and 65 years.
* BMI 18 - 32 kg/m².
* Positive skin prick test (wheal>4mm) with grasses pollen allergen extract.
* Specific IgE to grass pollen allergens by RAST (or equivalent test) ≥ class 2.
* Women of childbearing potential must be using a medically acceptable method of birth control and have a negative β-HCG pregnancy test result at screening and Day 1 predose. Male subjects must also agree to use the double barrier method of contraception during the study.
* In the opinion of the investigator, each subject will be able to understand verbal and written instructions and competent to follow these instructions.
* Subjects must read, understand, sign, and date the written informed consent form

Exclusion Criteria:

* Positive human immunodeficiency virus (HIV)-test, acute or chronic hepatitis B/C (except vaccination titer).
* Positive drug screen.
* Positive alcohol breath test.
* Known or suspected drug or alcohol abuse.
* History of clinically significant cardiovascular (especially heart failure or pulmonary insufficiency), pulmonary (except for asthma), hepatic, renal, gastrointestinal, hematologic, endocrine, dermatological, or metabolic disease within the last 2 years. A clinically significant disease is defined as a disease which, in the opinion of the investigator, may either put the subject at risk because of participation in the trial or a disease which may influence the results of the trial or the subject's eligibility to participate in the trial.
* Clinically significant abnormalities on pre-study physical examination, vital signs, electrocardiogram (ECG), or laboratory tests; acute illness within 7 days before the screening visit.
* History of allergy to all-season allergens and / or history of allergy to other seasonal allergens than grass pollen which might interfere with period of trial conduct
* History of a major psychiatric disorder such as schizophrenia, other psychotic symptomatology, major depressive disorder, or suicide attempt within the past 5 years; history of alcohol or drug abuse within the past year; history or evidence of a progressive central nervous system (CNS) disease, lesion, or encephalopathy.
* History of malignancy within the past 2 years; with the exception of basal cell carcinoma.
* Acute or subacute atopic dermatitis.
* Periodontitis, gingivitis, gingival bleeding or other mucosal disorders in the oral cavity or planned tooth extraction during the course of the study.
* Secondary changes of the reactive organs (e.g., emphysema, bronchiectasis).
* Auto-immune disease (e.g., of liver, kidney, thyroid, nervous system) rheumatoid diseases.
* Immunodeficiencies (e.g., by immunosuppressive agents).
* Therapy with β-blockers.
* Therapy with antihistamines less than three days prior to Day 1 .
* Therapy with corticosteroids (except hormonal contraceptives) four weeks prior to Day 1 (with the exception of local steroids, which must be terminated from three days prior to Day 1).
* Vaccinations in the last three months.
* Unable to comply with recommended therapy-free interval for specified medications prior to skin prick test.
* Current diseases with a pathogenesis interfering with the immune response and diseases for which medication has been given, which could influence the results of this study.
* Acute or chronic infection.
* Already undergone hyposensitization therapy with grass pollen allergens within the last three years.
* Use of MPL-containing products within the last 12 months or allergy / hypersensitivity to MPL.
* Pregnancy or breast-feeding.
* Use of any investigational drug or medical device within 30 days prior to the screening visit.
* A handicap that would prevent compliance with the study procedures or proper reporting of adverse events.
* Subjects who smoke more than 10 cigarettes a day
* Subjects unable to conduct nasal washes and comply with nasal challenge tests according to the instruction of the investigator
* Total flow during rhinomanometry with vehicle solution is more than 40% lower than total flow obtained with blank measurement (note: this exclusion criteria does not apply to the screening visit but to nasal challenge test performed on Day 1 predose)
* In the opinion of the investigator, unable to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events, | 18 weeks

SECONDARY OUTCOMES:
allergic reactions/symptomatology | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Timmer, MD, Principal Investigator — CRS Clinical Research Services Mannheim GmbH, Grenadierstraße 1, 68167 Mannheim, Germany
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany